CLINICAL TRIAL: NCT01887327
Title: A Phase 2b Multicenter, Single Dose, Randomized, Double Blind, Placebo-Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of Two Doses of Stannsoporfin in Combination With Phototherapy in Neonates
Brief Title: Stannsoporfin With Light Therapy for Newborn Babies With Jaundice
Acronym: JASMINE_204
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64,185-204
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Jaundice, Neonatal; Hyperbilirubinemia, Neonatal
Keywords: G6PD deficiency; Antibody (ABO) incompatibility; Coombs positive ABO/ rhesus factor (RH) incompatibility; Intensive phototherapy in neonates
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal; Glucosephosphate Dehydrogenase Deficiency | interventions — Phototherapy; tin mesoporphyrin; Drugs, Investigational; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants receive placebo and phototherapy
  Interventions: Procedure: Phototherapy; Drug: Placebo
- Stannsoporfin 3.0 mg/kg (Experimental): Participants receive stannsoporfin (3.0 mg/kg) and phototherapy
  Interventions: Procedure: Phototherapy; Drug: Stannsoporfin
- Stannsoporfin 4.5 mg/kg (Experimental): Participants receive stannsoporfin (4.5 mg/kg) and phototherapy
  Interventions: Procedure: Phototherapy; Drug: Stannsoporfin

INTERVENTIONS:
Procedure: Phototherapy — Phototherapy starts within 30 minutes before or after injection
  Other Names: Light therapy
Drug: Stannsoporfin — Stannsoporfin (3.0 or 4.5 mg/kg) administered by intramuscular (IM) injection (a shot in the muscle)
  Other Names: Experimental drug
  Arms: Stannsoporfin 3.0 mg/kg; Stannsoporfin 4.5 mg/kg
Drug: Placebo — Matching placebo administered by IM injection
  Other Names: Matching placebo; Saline
  Arms: Placebo

SUMMARY:
It is normal for red blood cells to die, even in newborn babies. The waste from that is called bilirubin. The liver clears bilirubin out of the body.

Some babies are born with illness that makes red blood cells die too fast, so the liver is not strong enough to keep up with it.

The yellowish color in eyes or skin means there is too much bilirubin in the body. It can be dangerous if a baby's bilirubin gets too high.

Special lights are put on jaundiced babies (called phototherapy) to help the liver get rid of bilirubin.

This study tests an experimental drug to see if it can help the liver even more, by safely cutting down the amount of bilirubin the body is making in the first place.

DETAILED DESCRIPTION:
Participants randomized (1:1:1) to treatment groups will be term or near-term infants with isoimmune hemolytic disease or glucose-6-phosphate dehydrogenase (G6PD) deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Term and near term infants ≥35 and ≤ 43 weeks gestational age (GA), age 0-48 hours with antibody (ABO) or rhesus factor (Rh) incompatibility (anti C, c, D, E or e) who are Coombs positive, or age 0-72 hours with G6PD deficiency
2. Parental or guardian consent
3. Birth weight ≥ 2500 grams
4. At or above the age-specific threshold for initiating phototherapy (PT) per the American Academy of Pediatrics (AAP) guidelines based on measurement of total serum bilirubin (TSB)
5. Parents agree to observe light precautions for 10 days post treatment

Exclusion Criteria:

1. Elevated direct bilirubin ≥2 mg/dL, OR > 20% of the total serum bilirubin
2. Alanine aminotransferase (ALT) > 2 times the upper limit of normal (ULN) and/or aspartate aminotransferase (AST) > 3 times ULN
3. Abnormal renal function defined as creatinine and/or blood urea nitrogen >2 times the ULN
4. Any other clinically significant abnormalities on screening laboratory evaluation [including electrocardiogram (ECG)] that in the opinion of the investigator makes the patient unsuitable for the clinical trial
5. Apgar score ≤6 at age 5 minutes
6. An unexplained existing rash or skin erythema
7. Prior exposure to PT
8. Clinical suggestion of neonatal thyroid disease or current uncontrolled thyroid disease in the mother (maternal Hashimoto's disease is not exclusionary)
9. Cardio-respiratory distress, defined as a respiratory rate >60 breaths per minute at time of enrollment
10. Any abnormal auditory or ophthalmologic findings on screening physical exam
11. Treatment or need for treatment in the neonate with medications that are photoreactive or may prolong the QT interval (erythromycin ointment for eye prophylaxis is permitted), or family history of Long QT syndrome
12. Known porphyrias or risk factors for porphyrias, including family history
13. A maternal history of systemic lupus erythematosus
14. Maternal use of phenobarbital 30 days before, or after delivery, if breast-feeding
15. Maternal current drug or alcohol abuse, or maternal history of drug or alcohol abuse that, in the opinion of the Investigator, would not make the patient a suitable candidate for participation in the clinical trial
16. Significant congenital anomalies or infections
17. Risk of requiring surgery or exposure to operating room (OR) lights in the first 2 weeks of life
18. Persistent hypoglycemia (blood glucose <40 mg/dL)
19. Temperature instability defined as temperature consistently (3 consecutive times) <36 degrees centigrade (ºC) and/or >37.5 degrees centigrade (ºC) axillary
20. Use of intravenous immunoglobulin (IVIg) or albumin prior to study drug administration
21. Post-delivery treatment with medications that are known or suspected to displace bilirubin from albumin (e.g., ceftriaxone or sulfa-based antibiotics)
22. Use of photosensitizing drugs or agents
23. Unwillingness of parents/guardians to adhere to recommendations regarding light precautions
24. Exposure to any investigational medications or devices after delivery, or participation in another clinical trial while participating in this trial
25. Any other concurrent medical condition, which in the opinion of the Investigator, makes the patient unsuitable for the clinical trial

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2016-03-22 (Actual); Study Completion 2016-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company
Locations (18):
- United States (18):
  - Arrowhead Regional Medical Center, Colton, California
  - University of California San Diego Medical Center, San Diego, California
  - University of CA, San Francisco, San Francisco, California
  - Univ Florida Hospital, Jacksonville, Florida
  - Kosair Children's Hospital, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Univ Med Ctr of Southern Nevada, Las Vegas, Nevada
  - Rutgers University Hospital, Newark, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Stoney Brook Univ Hospital, Stony Brook, New York
  - WakeMed Health and Hospitals, Raleigh, North Carolina
  - Toledo Children's Hospital, Toledo, Ohio
  - Hahnemann University Hospital/St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical Univ of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - JPS Health Network, Fort Worth, Texas
  - Univ Texas Medical Branch, Galveston, Texas
  - Children's Hospital of Richmond at VCU, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- 3.0 mg/kg Stannsoporfin: Participants receive 3.0 mg/kg Stannsoporfin and phototherapy
- 4.5 mg/kg Stannsoporfin: Participants receive 4.5 mg/kg stannsoporfin and phototherapy
Period: Overall Study
Arm/Group | 3.0 mg/kg Stannsoporfin | 4.5 mg/kg Stannsoporfin | Placebo
Started | 30 | 31 | 30
Completed | 29 | 27 | 27
Not Completed | 1 | 4 | 3

BASELINE CHARACTERISTICS:
Population: ITT Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.0 mg/kg Stannsoporfin | 4.5 mg/kg Stannsoporfin | Placebo | Total
Number analyzed (Participants) | 30 | 31 | 30 | 91
Age, Continuous [Mean (Standard Deviation); unit: Hour] | 21.66 (11.417) | 24.05 (11.020) | 25.92 (12.361) | 23.88 (11.608)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 13 | 43
  Male | 15 | 16 | 17 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 15 | 31
  Not Hispanic or Latino | 23 | 22 | 15 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 13 | 9 | 38
  White | 9 | 13 | 12 | 34
  More than one race | 4 | 5 | 8 | 17
  Unknown or Not Reported | 1 | 0 | 0 | 1
Age at Qualifying TSB [Count of Participants; unit: Participants]
  Less than or equal to 12 h | 13 | 12 | 10 | 35
  Greater than 12 h to Less than or equal to 24 h | 11 | 8 | 7 | 26
  Greater than 24 h to Less than or equal to 32 h | 3 | 7 | 7 | 17
  Greater than 32 h to Less than or equal to 40 h | 1 | 2 | 3 | 6
  Greater than 40 h | 2 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Total Serum Bilirubin (mg/dL)
Description: Total serum bilirubin (TSB) was measured at baseline (the measure that qualified the baby for inclusion) and at 48 hours after treatment. If a baby was discharged before 48 hours, the last measurement before discharge was used [last observation carried forward (LOCF)].
Time Frame: Baseline, 48 hours post-treatment
Population: Intention to treat (ITT) analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 3.0 mg/kg Stannsoporfin | 4.5 mg/kg Stannsoporfin | Placebo
Number analyzed (Participants) | 30 | 31 | 30
mg/dL
  Baseline | 9.82 (2.641) | 9.97 (2.967) | 9.92 (2.211)
  48 hours post-treatment | 8.48 (1.973) | 8.86 (2.142) | 11.67 (2.337)
Statistical Analysis 1: Comparison: 3.0 mg/kg Stannsoporfin vs Placebo; Test type: Other; p = 0.0000021, LS Mean Difference vs Placebo; LS Mean Difference vs Placebo = -31.64, 95% CI 2-sided [-44.000 to -19.283]
Statistical Analysis 2: Comparison: 4.5 mg/kg Stannsoporfin vs Placebo; Test type: Other; p = 0.0000260, LS Mean Difference vs Placebo; LS Mean Difference vs Placebo = -27.40, 95% CI 2-sided [-39.657 to -15.142]

2. Secondary Outcome: Time (Hour) at Which TSB First Crosses at or Below the Defined Age-specific Threshold for 54-hours Post-treatment (PT)
Description: The hour that 50% of babies in the group (median) first crosses at or below the defined 54-hour threshold for the baby's age
Time Frame: within 54 hours
Population: ITT Analysis Set minus 2 participants who received placebo and did not reach the defined threshold for their age within 54 hours
Measure: Median (Full Range); unit: hours
Arm/Group | 3.0 mg/kg Stannsoporfin | 4.5 mg/kg Stannsoporfin | Placebo
Number analyzed (Participants) | 30 | 31 | 28
hours | 11.8 [-3.7 to 53.6] | 10.6 [-5.5 to 28.5] | 20.9 [-4.4 to 54.0]

3. Secondary Outcome: Number of Participants With Phototherapy (PT) Failure
Description: PT failure was defined by any of the following:
  * re-start of PT within 6 hours after stopping
  * re-hospitalization for hyperbilirubinaemia
  * use of intravenous immunoglobulin (IVIg)
  * need for an exchange transfusion
Time Frame: within 30 days after discharge
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | 3.0 mg/kg Stannsoporfin | 4.5 mg/kg Stannsoporfin | Placebo
Number analyzed (Participants) | 30 | 31 | 30
Participants
  PT failure Occurred | 3 | 1 | 8
  Did not occur | 27 | 30 | 22

4. Secondary Outcome: Number of Participants With Rebound Hyperbilirubinemia
Description: Rebound hyperbilirubinaemia was defined as an increase in TSB above the age-specific threshold for initiating phototherapy, following the discontinuation of the initial phototherapy.
Time Frame: within 54 hours
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | 3.0 mg/kg Stannsoporfin | 4.5 mg/kg Stannsoporfin | Placebo
Number analyzed (Participants) | 30 | 31 | 30
Participants
  Occurred | 0 | 1 | 3
  Did not occur | 30 | 30 | 27

ADVERSE EVENTS:
Time Frame: within 30 Days
Description: Only treatment-emergent adverse events are reported. Treatment-emergent adverse events are those that started or got worse after treatment. Participants with multiple occurrences of a preferred term were counted only once for that preferred term.
Groups:
- 4.5mg/kg Stannsoporfin: Participants receive 4.5mg/kg stannsoporfin and phototherapy
Arm/Group | 3.0 mg/kg Stannsoporfin | 4.5mg/kg Stannsoporfin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 5/30 | 4/31 | 6/30
Other Adverse Events (participants affected / at risk) | 28/30 | 21/31 | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3.0 mg/kg Stannsoporfin (N=30) | 4.5mg/kg Stannsoporfin (N=31) | Placebo (N=30)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 3
ABO incompatibility (Immune system disorders) | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Hematocrit decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Medical observation (Investigations) | 2 | 0 | 0
Reticulocyte count increased (Investigations) | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3.0 mg/kg Stannsoporfin (N=30) | 4.5mg/kg Stannsoporfin (N=31) | Placebo (N=30)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Congenital naevus (Congenital, familial and genetic disorders) | 0 | 2 | 2
Conjucunctival Hemorrhage (Eye disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 4 | 1 | 0
Fat Tissue Increased (General disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 3
Bacterial Sepsis (Infections and infestations) | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 2
Cardiac murmur (Investigations) | 5 | 4 | 4
Gamma-glutamyl transferase increased (Investigations) | 2 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 2 | 1
Haemoglobin decreased (Investigations) | 2 | 1 | 1
Medical observation (Investigations) | 2 | 0 | 0
Reticulocyte count increased (Investigations) | 2 | 3 | 1
Abnormal Loss Of Weight (Metabolism and nutrition disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acne infantile (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 5 | 5 | 0
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Milia (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Platelet Toxicity (Blood and lymphatic system disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular Hypertrophy (Cardiac disorders) | 1 | 0 | 0
Ankyloglossia Congenital (Congenital, familial and genetic disorders) | 1 | 0 | 0
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 | 0 | 0
Dacryostenosis Congenital (Congenital, familial and genetic disorders) | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0
Patent Ductus Arteriosus (Congenital, familial and genetic disorders) | 1 | 0 | 0
Middle Ear Effusion (Ear and labyrinth disorders) | 0 | 1 | 0
Eye Discharge (Eye disorders) | 1 | 0 | 0
Ocular Icterus (Eye disorders) | 0 | 0 | 1
Retinal Haemorrhage (Eye disorders) | 0 | 1 | 0
Strabismus (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Infantile Colic (Gastrointestinal disorders) | 1 | 0 | 0
Infantile Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Injection Site Erythema (General disorders) | 0 | 1 | 0
Abo Incompatibility (Immune system disorders) | 0 | 0 | 1
Candida Nappy Rash (Infections and infestations) | 1 | 0 | 0
Fungal Infection (Infections and infestations) | 0 | 1 | 0
Meningitis Viral (Infections and infestations) | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Skin Candida (Infections and infestations) | 1 | 0 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 1 | 0
Bilirubin Conjugated Increased (Investigations) | 1 | 0 | 0
Blood Bicarbonate Decreased (Investigations) | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0
Carbon Dioxide Decreased (Investigations) | 0 | 0 | 1
Haematocrit Abnormal (Investigations) | 1 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1 | 0
Red Blood Cell Count Decreased (Investigations) | 0 | 1 | 0
Respiratory Syncytial Virus Test Positive (Investigations) | 1 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1 | 0
Feeding Intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Umbilical Granuloma (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Jaundice Neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Penile Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Neonatal Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cafe Au Lait Spots (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Generalised Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Melanosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash Neonatal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Sensitisation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Transient Neonatal Pustular Melanosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No